CLINICAL TRIAL: NCT05275023
Title: A Phase 2 Open-label Trial to Evaluate Safety, Efficacy, Tolerability, and Pharmacodynamics of a Combination of JNJ-73763989, Nucleos(t)Ide Analogs, and a PD-1 Inhibitor in Chronic Hepatitis B Patients
Brief Title: An Efficacy and Safety Study of a Combination of JNJ-73763989, Nucleos(t)Ide Analogs (NA), and a Programmed Cell Death Protein Receptor-1 (PD-1) Inhibitor in Chronic Hepatitis B Participants
Acronym: OCTOPUS-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109161; 73763989PAHPB2008 (Other: Janssen Research & Development, LLC); 2021-005132-33 (EudraCT Number)
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Immune Checkpoint Inhibitors; Tenofovir; tenofovir alafenamide; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1: JNJ-73763989 + PD-1 Inhibitor + Nucleos(t)ide analog (NA) (Experimental): Participants will receive JNJ-73763989 subcutaneous (SC) injections and single dose of programmed cell death protein receptor-1 (PD-1) inhibitor as intravenous (IV) infusion. Participants will also receive background treatment with NA (either tenofovir disoproxil, tenofovir alafenamide [TAF] or entecavir [ETV]).
  Interventions: Drug: JNJ-73763989; Drug: PD-1 inhibitor; Drug: Tenofovir Disoproxil; Drug: Tenofovir Alafenamide; Drug: Entecavir
- Arm 2: JNJ-73763989 + PD-1 Inhibitor + NA (Experimental): Participants will receive JNJ-73763989 SC injections and multiple doses of PD-1 inhibitor as IV infusion. Participants will also receive background treatment with NA (either tenofovir disoproxil, TAF or ETV).
  Interventions: Drug: JNJ-73763989; Drug: PD-1 inhibitor; Drug: Tenofovir Disoproxil; Drug: Tenofovir Alafenamide; Drug: Entecavir

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered subcutaneously.
  Other Names: JNJ-3989
Drug: PD-1 inhibitor — PD-1 inhibitor will be administered as IV infusion.
Drug: Tenofovir Disoproxil — Tenofovir disoproxil film-coated tablets will be administered orally.
Drug: Tenofovir Alafenamide — TAF film-coated tablets will be administered orally.
Drug: Entecavir — ETV film-coated tablets will be administered orally.

SUMMARY:
The purpose of this study is to evaluate efficacy of the study intervention, based on hepatitis B surface antigen (HBsAg) levels at follow-up (FU) Week 24.

DETAILED DESCRIPTION:
JNJ-73763989 (JNJ-3989) is a small interfering ribonucleic acid (siRNA) targeting all hepatitis B virus (HBV) messenger ribonucleic acid (mRNAs). The programmed cell death protein receptor-1 (PD-1) inhibitor aims at preventing the interaction of PD-1 with its ligands. The purpose of this study to determine whether at least one of the combination regimens of JNJ-3989 + PD-1 inhibitor + Nucleos(t)ide analog (NA) is more efficacious than JNJ-3989 + NA treatment. This study will be conducted in 3 periods: screening period, treatment period and follow-up (FU) period. Safety assessments will include adverse events (AEs), serious AEs, clinical safety laboratory tests, electrocardiograms (ECGs), vital signs, and physical examinations. Total duration of individual participation will be up to 78 weeks (including screening period).

ELIGIBILITY:
Inclusion Criteria:

* Participants must have chronic hepatitis B virus (HBV) infection
* Participants must have fibroscan liver stiffness measurement less than or equal to (<=) 9.0 kilopascal (kPa) or a liver biopsy result classified as metavir F0-F2

Exclusion Criteria:

* Participants with evidence of hepatitis A virus infection (hepatitis A antibody immunoglobulin IgM), hepatitis C virus (HCV) infection (HCV antibody), hepatitis D virus (HDV) infection (HDV antibody), hepatitis E virus (HEV) infection (hepatitis E antibody IgM), or human immunodeficiency virus type 1 (HIV-1) or human immunodeficiency virus type 2 (HIV-2) infection (laboratory confirmed) at screening
* History or evidence of clinical signs or symptoms of hepatic decompensation, including but not limited to portal hypertension, ascites, hepatic encephalopathy, esophageal varices
* Participants with history or signs of cirrhosis or portal hypertension or signs of hepatocellular carcinoma (HCC) or clinically relevant renal abnormalities
* Participants with personal/familial history/indicative of immune-mediated disease risk

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (26):
- Toronto General Hospital, Toronto, Ontario, Canada
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - IKEM, Prague
- France (4):
  - Hopital Beaujon, Clichy
  - Hopital Saint Joseph, Marseille
  - Chu Rennes Hopital Pontchaillou, Rennes
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Italy (3):
  - Fondazione IRCCS Ca Granda Ospedale Policlinico Di Milano, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Universita degli Studi di Roma 'La Sapienza' - Umberto I Policlinico di Roma, Rome
- Spain (4):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Pta. de Hierro Majadahonda, Madrid
  - Hosp. Montecelo, Pontevedra
  - Hosp. Gral. Univ. Valencia, Valencia
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (5):
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Karadeniz Teknik University Medical Faculty, Trabzon
- United Kingdom (3):
  - Glasgow Royal Infirmary, Glasgow
  - Kings College Hospital, London
  - Imperial College London and Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + Nucleos(t)Ide Analog (NA): In intervention phase (IP), participants received a loading dose of JNJ-3989 200 milligrams (mg) as subcutaneous (SC) injection once weekly (QW) for first 4 weeks starting from Week 0 up to Week 3 followed by single dose once every 4 weeks (Q4W) from Week 4 up to Week 24. At Week 16, participants received a single dose of nivolumab 0.3 milligrams per kilogram (mg/kg) as intravenous (IV) infusion. Participants also received NA (either tenofovir disoproxil 245 mg or tenofovir alafenamide [TAF] 25 mg or entecavir [ETV] 0.5 mg) tablet orally once daily (QD) from Week 0 up to Week 24. After Week 24, participants were followed up for safety for 48 weeks during which they continued to receive NA (tenofovir disoproxil 245 mg or TAF 25 mg or ETV 0.5 mg) tablet orally QD up to follow up (FU) Week 48 (up to Week 72).
- JNJ-3989 + Nivolumab (3 Infusions) + NA: In IP, participants received a loading dose of JNJ-3989 200 mg as SC injection QW for first 4 weeks starting from Week 0 up to Week 3 followed by single dose Q4W from Week 4 up to Week 24. At Weeks 16, 20 and 24, participants received of nivolumab 0.3 mg/kg as IV infusion. Participants also received NA (either tenofovir disoproxil 245 mg or TAF 25 mg or ETV 0.5 mg) tablet orally QD from Week 0 up to Week 24. After Week 24, participants were followed up for safety for 48 weeks during which they continued to receive NA (tenofovir disoproxil 245 mg or TAF 25 mg or ETV 0.5 mg) tablet orally QD up to FU Week 48 (up to Week 72).
Period: Intervention Phase: Week 0 to Week 24
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + Nucleos(t)Ide Analog (NA) | JNJ-3989 + Nivolumab (3 Infusions) + NA
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0
Period: FU Phase: FU Week 1 to FU Week 48
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + Nucleos(t)Ide Analog (NA) | JNJ-3989 + Nivolumab (3 Infusions) + NA
Started | 18 | 19
Completed | 18 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA: In intervention phase (IP), participants received a loading dose of JNJ-3989 200 milligrams (mg) as subcutaneous (SC) injection once weekly (QW) for first 4 weeks starting from Week 0 up to Week 3 followed by single dose once every 4 weeks (Q4W) from Week 4 up to Week 24. At Week 16, participants received a single dose of nivolumab 0.3 mg/kg as IV infusion. Participants also received NA (either tenofovir disoproxil 245 mg or tenofovir alafenamide [TAF] 25 mg or entecavir [ETV] 0.5 mg) tablet orally once daily (QD) from Week 0 up to Week 24. After Week 24, participants were followed up for safety for 48 weeks during which they continued to receive NA (tenofovir disoproxil 245 mg or TAF 25 mg or ETV 0.5 mg) tablet orally QD up to FU Week 48 (up to Week 72).
- Total: Total of all reporting groups
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 5
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  CANADA | 3 | 2 | 5
  FRANCE | 0 | 2 | 2
  ITALY | 3 | 2 | 5
  SPAIN | 2 | 5 | 7
  TAIWAN | 3 | 4 | 7
  TURKEY | 6 | 3 | 9
  UNITED KINGDOM | 1 | 1 | 2
AgeContinuous [Mean (Standard Deviation); unit: years] | 40.7 (7.75) | 47.9 (5.05) | 44.4 (7.38)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Hepatitis B Surface Antigen (HBsAg) Seroclearance at Follow-up (FU) Week 24
Description: Percentage of participants who achieved HBsAg seroclearance at FU Week 24 were reported. Seroclearance of HBsAg was defined as a (quantitative) HBsAg level less than (<) lower limit of quantification (LLOQ) (0.05 international unit per milliliters [IU/mL]).
Time Frame: At FU Week 24
Population: Full analysis set (FAS) included all participants who were randomly assigned to an intervention arm in this intervention-specific appendix (ISA) and received at least 1 dose of study intervention within this ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants | 0 | 0

2. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs) of Special Interest
Description: An AE was any untoward medical occurrence in a participant participating in a clinical study that does not necessarily had a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after the initial administration of study intervention was considered to be treatment emergent. AEs of interest were significant AEs that are judged to be of special interest because of clinical importance, known class effects or based on nonclinical signals.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP | 11.1 | 5.3
  FU Phase | 0 | 5.3

3. Secondary Outcome: Number of Participants With TEAEs by Severity
Description: Number of participants with TEAEs by severity were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that did not necessarily had a causal relationship with the pharmaceutical/biological agent under study. Any AE occurring at or after the initial administration of study intervention was considered to be treatment emergent. Severity of AE were graded by using Division of Acquired Immunodeficiency Syndrome (DAIDS) grading scale that ranges from Grade 1 to Grade 5. Grade 1 indicates a mild event, Grade 2 indicates a moderate event, Grade 3 indicates a severe event, Grade 4 indicated a potentially life-threatening event, Grade 5 indicated death.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Participants
  IP: Grade 1 | 5 | 7
  IP: Grade 2 | 1 | 5
  IP: Grade 3 | 0 | 0
  IP: Grade 4 | 0 | 0
  IP: Grade 5 | 0 | 0
  FU Phase: Grade 1 | 7 | 6
  FU Phase: Grade 2 | 1 | 2
  FU Phase: Grade 3 | 0 | 0
  FU Phase: Grade 4 | 0 | 0
  FU Phase: Grade 5 | 0 | 0

4. Secondary Outcome: Number of Participants With Immune Related TEAEs
Description: Number of participants with immune related TEAEs were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that did not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. Any AE occurring at or after the initial administration of study intervention was considered to be treatment emergent. Immune-related AEs (irAEs) were alanine aminotransferase/alanine aminotransferase (ALT/AST) elevations including immune-related hepatic AEs, infusion-related reaction (IRRs) and other irAEs (including gastrointestinal AEs, neurological AEs, pulmonary AEs, renal AEs, endocrinopathies, rash, uveitis and visual complaints, lipase/amylase elevations, and infection), hematological abnormalities and injection site reactions.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Participants
  IP | 0 | 0
  FU Phase | 0 | 1

5. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Number of participants with abnormalities in vital signs measurements (including pulse rate: abnormally low: less than or equal to [<=] 45 beats per minute [bpm], abnormally high: greater than or equal to [>=] 120 bpm; diastolic blood pressure [BP]: abnormally low: <=50 millimeters of mercury [mmHg], mild: >90 to <100 mmHg, moderate: >=100 to <110 mmHg, and severe: >=110 mmHg; systolic BP: abnormally low: <=90 mmHg, mild: >140 to <160 mmHg, moderate: >=160 to <180 mmHg, and severe: >=180 mmHg) were reported.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Participants
  IP: Pulse: Abnormally Low | 0 | 0
  IP: Pulse: Abnormally High | 0 | 0
  IP: Diastolic BP: Abnormally Low | 0 | 0
  IP: Diastolic BP: Mild | 0 | 1
  IP: Diastolic BP: Moderate | 0 | 1
  IP: Diastolic BP: Severe | 0 | 1
  IP: Systolic BP: Abnormally low | 2 | 2
  IP: Systolic BP: Mild | 2 | 1
  IP: Systolic BP: Moderate | 0 | 1
  IP: Systolic BP: Severe | 0 | 0
  FU Phase: Pulse: Abnormally low | 0 | 0
  FU Phase: Pulse: Abnormally high | 0 | 0
  FU Phase: Diastolic BP: Abnormally low | 0 | 1
  FU Phase: Diastolic BP: Mild | 1 | 1
  FU Phase: Diastolic BP: Moderate | 0 | 1
  FU Phase: Diastolic BP: Severe | 0 | 0
  FU Phase: Systolic BP: Abnormally low | 0 | 0
  FU Phase: Systolic BP: Mild | 2 | 2
  FU Phase: Systolic BP: Moderate | 0 | 0
  FU Phase: Systolic BP: Severe | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormalities in 12-lead Electrocardiogram (ECGs)
Description: Number of participants with abnormalities in 12-lead ECGs: heart rate (abnormally low: <45 beats per minute [bpm], abnormally high: greater than or equal [>=] 120 bpm), PR interval (abnormally high: greater than [>] 220 millisecond [msec]), QRS interval (abnormally high: >=120 msec), QTc interval Fridericia (Borderline prolonged QT: 450< QTc <=480 msec; Prolonged QT: 480 < QTc <=500; Pathologically prolonged QT: QTc >500) were reported.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA. Here, 'n' (number analyzed) refers to number of participants evaluable at specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Participants
  IP: Heart rate: Abnormally low | 0 | 0
  IP: Heart rate: Abnormally high | 0 | 0
  IP: PR interval: Abnormally high | 1 | 0
  IP: QRS interval: Abnormally high | 0 | 0
  IP: QTc interval: Borderline prolonged QT | 0 | 1
  IP: QTc interval: prolonged QT | 0 | 0
  IP: QTc interval: Pathologically prolonged QT | 0 | 0
  FU Phase: Heart rate: Abnormally low: number analyzed (Participants) | 18 | 18
  FU Phase: Heart rate: Abnormally low | 0 | 0
  FU Phase: Heart rate: Abnormally high: number analyzed (Participants) | 18 | 18
  FU Phase: Heart rate: Abnormally high | 0 | 0
  FU Phase: PR interval: Abnormally high: number analyzed (Participants) | 18 | 18
  FU Phase: PR interval: Abnormally high | 0 | 0
  FU Phase: QRS interval: Abnormally high: number analyzed (Participants) | 18 | 18
  FU Phase: QRS interval: Abnormally high | 0 | 0
  FU Phase: QTc interval Borderline prolonged QT: number analyzed (Participants) | 18 | 18
  FU Phase: QTc interval Borderline prolonged QT | 0 | 1
  FU Phase: QTc interval: prolonged QT: number analyzed (Participants) | 18 | 18
  FU Phase: QTc interval: prolonged QT | 0 | 0
  FU Phase:QTc interval: Pathologically prolonged QT: number analyzed (Participants) | 18 | 18
  FU Phase:QTc interval: Pathologically prolonged QT | 0 | 0

7. Secondary Outcome: Number of Participants With Abnormalities in Physical Examinations
Description: Number of participants with abnormalities in physical examinations were reported.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Participants
  IP | 0 | 2
  FU Phase | 2 | 1

8. Secondary Outcome: Percentage of Participants With Abnormalities in Clinical Laboratory Parameters: Hematology
Description: Percentage of participants with abnormalities in hematology parameters (including basophils/Leukocytes high, erythrocytes mean corpuscular volume high, erythrocytes high and low, lymphocytes/leukocytes high and low, monocytes/leukocytes high and low, neutrophils, segmented+band form high and low, reticulocytes/erythrocytes high and low, basophils/leukocytes, eosinophils/leukocytes high, erythrocyte mean corpuscular hemoglobin low, reticulocytes/erythrocytes high and low, lymphocytes atypical/leukocytes high, lymphocytes atypical high, hematocrit high, monocytes low and high) were reported. Abnormalities with at least 1 participant is included. Low and high categorization depend on investigator's discretion.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA. Here, 'n' (number analyzed) refers to number of participants evaluable at specified parameter. n=0 indicates that there was no evaluable participant for specified parameter.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + Nucleos(t)Ide Analog (NA) | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP: Basophils/Leukocytes: High | 11.1 | 42.1
  IP: Erythrocytes Mean Corpuscular Volume: High | 16.7 | 0
  IP: Erythrocytes: Low | 16.7 | 26.3
  IP: Erythrocytes: High | 0 | 5.3
  IP: Lymphocytes/Leukocytes: Low | 0 | 5.3
  IP: Lymphocytes/Leukocytes: High | 11.1 | 5.3
  IP: Monocytes/Leukocytes: Low | 0 | 5.3
  IP: Monocytes/Leukocytes: High | 0 | 5.3
  IP: Neutrophils, Segmented+Band Form: Low | 22.2 | 26.3
  IP: Neutrophils, Segmented+Band Form: High | 11.1 | 10.5
  IP: Reticulocytes/Erythrocytes: Low | 0 | 10.5
  IP: Reticulocytes/Erythrocytes: High | 0 | 10.5
  FU Phase: Basophils/Leukocytes: High | 11.1 | 5.3
  FU Phase: Eosinophils/Leukocytes: High | 0 | 15.8
  FU Phase: Erythrocyte Mean Corpuscular Hemoglobin: Low | 5.6 | 0
  FU Phase: Erythrocyte Mean Corpuscular Volume: High | 27.8 | 15.8
  FU Phase: Erythrocyte: Low | 11.1 | 21.1
  FU Phase: Erythrocyte: High | 0 | 5.3
  FU Phase: Lymphocytes/Leukocytes: Low | 11.1 | 5.3
  FU Phase: Lymphocytes/Leukocytes: High | 22.2 | 5.3
  FU Phase: Monocytes/Leukocytes: Low | 0 | 10.5
  FU Phase: Monocytes/Leukocytes: High | 5.6 | 15.8
  FU Phase: Neutrophils, Segmented + Band Form: Low | 38.9 | 31.6
  FU Phase: Neutrophils, Segmented + Band Form: High | 11.1 | 0
  FU Phase: Reticulocytes/Erythrocytes: Low | 16.7 | 42.1
  FU Phase: Reticulocytes/Erythrocytes: High | 0 | 5.3
  FU Phase: Lymphocytes Atypical/Leukocytes: High: number analyzed (Participants) | 0 | 1
  FU Phase: Lymphocytes Atypical/Leukocytes: High |  | 100
  FU Phase: Lymphocytes Atypical: High: number analyzed (Participants) | 0 | 1
  FU Phase: Lymphocytes Atypical: High |  | 100
  FU Phase: Hematocrit: High | 5.6 | 0
  FU Phase: Monocytes: Low | 5.6 | 10.5
  FU Phase: Monocytes: High | 5.6 | 0

9. Secondary Outcome: Number of Participants With Abnormalities in Clinical Laboratory Parameters: Clinical Chemistry
Description: Number of participants with abnormalities in clinical chemistry parameters (including C reactive protein high, cystatin C low and high, gamma glutamyl transferase low, high density lipoprotein [HDL] cholesterol low and high, indirect bilirubin high, lactate dehydrogenase high, protein high, thyrotropin low and high, free thyroxine high, free triiodothyronine low and high, and urea nitrogen high) were reported. Abnormalities with at least 1 participant is included. Low and high categorization depend on investigator's discretion.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Participants
  IP: C Reactive Protein: High | 3 | 2
  IP: Cystatin C: Low | 2 | 1
  IP: Cystatin C: High | 1 | 1
  IP: Gamma Glutamyl Transferase: Low | 4 | 4
  IP: HDL Cholesterol: Low | 6 | 3
  IP: HDL Cholesterol: High | 3 | 4
  IP: Indirect Bilirubin: High: number analyzed (Participants) | 18 | 17
  IP: Indirect Bilirubin: High | 1 | 0
  IP: Lactate Dehydrogenase: High | 2 | 2
  IP: Protein: High | 1 | 0
  IP: Thyrotropin: Low | 2 | 0
  IP: Thyrotropin: High | 1 | 0
  IP: Free Thyroxine: High | 3 | 1
  IP: Triiodothyronine, Free: Low | 0 | 1
  IP: Triiodothyronine, Free: High | 5 | 4
  IP: Urea Nitrogen: High | 1 | 2
  FU Phase: C Reactive Protein: High | 2 | 0
  FU Phase: Chloride: Low | 0 | 1
  FU Phase: Cystatin C: Low | 1 | 0
  FU Phase: Cystatin C: High | 2 | 3
  FU Phase: Gamma Glutamyl Transferase: Low | 0 | 1
  FU Phase: HDL Cholesterol: Low | 6 | 2
  FU Phase: HDL Cholesterol: High | 2 | 4
  FU Phase: Indirect Bilirubin: High: number analyzed (Participants) | 17 | 18
  FU Phase: Indirect Bilirubin: High | 1 | 0
  FU Phase: Lactate Dehydrogenase: High | 2 | 2
  FU Phase: Protein: High | 1 | 1
  FU Phase: Thyrotropin: Low | 1 | 0
  FU Phase: Thyrotropin: High | 1 | 1
  FU Phase: Free Thyroxine: Low | 1 | 1
  FU Phase: Free Thyroxine: High | 2 | 0
  FU Phase: Free Triiodothyronine: High | 6 | 3
  FU Phase: Urea Nitrogen: High | 1 | 1

10. Secondary Outcome: Number of Participants With Abnormalities in Clinical Laboratory Parameters: Urinalysis
Description: Number of participants with abnormalities in clinical laboratory parameters (including specific gravity high and urine hyaline casts high) were reported. Abnormalities with at least 1 participant is included. Low and high categorization depend on investigator's discretion.
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: Safety analysis set included all participants who received at least 1 dose of study intervention within this ISA. Here, N (number of participants analyzed) signifies number of participants analyzed for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 9 | 11
Participants
  IP: Specific Gravity: High | 2 | 0
  IP: Urine Hyaline Casts: High: number analyzed (Participants) | 1 | 1
  IP: Urine Hyaline Casts: High | 1 | 1
  FU Phase: Specific Gravity: High: number analyzed (Participants) | 8 | 7
  FU Phase: Specific Gravity: High | 1 | 1
  FU Phase: Urine Hyaline Casts: High: number analyzed (Participants) | 2 | 2
  FU Phase: Urine Hyaline Casts: High | 2 | 2

11. Secondary Outcome: Change From Baseline in Hepatitis B Surface Antigen (HBsAg) Levels
Description: Change from baseline in HBsAg levels were reported. International units per milliliters=IU/mL. End of Study Intervention (EOSI) was the last post-baseline visit in study intervention period. End of study (EOS) was the last visit in the study.
Time Frame: IP: Baseline, Weeks 1, 2, 3, 4, 8, 12, 16, 20, and End of Study Intervention (EOSI; Week 24); FU Phase: FU Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, and EOS (last visit at FU Week 48)
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoints.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
log10 IU/mL
  IP: Baseline | 3.25 (0.472) | 3.14 (0.542)
  IP: Week 1 | -0.19 (0.185) | -0.17 (0.135)
  IP: Week 2 | -0.26 (0.293) | -0.31 (0.330)
  IP: Week 3 | -0.34 (0.335) | -0.44 (0.405)
  IP: Week 4 | -0.40 (0.400) | -0.52 (0.525)
  IP: Week 8 | -0.80 (0.576) | -0.87 (0.695)
  IP: Week 12 | -1.32 (0.513) | -1.41 (0.687)
  IP: Week 16 | -1.77 (0.361) | -1.84 (0.548)
  IP: Week 20 | -1.97 (0.376) | -2.07 (0.549)
  IP: EOSI (Week 24) | -2.01 (0.385) | -2.10 (0.563)
  FU Phase: Week 4: number analyzed (Participants) | 6 | 7
  FU Phase: Week 4 | -1.93 (0.515) | -1.98 (0.590)
  FU Phase: Week 8 | -1.99 (0.417) | -2.12 (0.613)
  FU Phase: Week 12: number analyzed (Participants) | 17 | 16
  FU Phase: Week 12 | -1.93 (0.393) | -1.99 (0.574)
  FU Phase: Week 16 | -1.85 (0.420) | -2.01 (0.648)
  FU Phase: Week 20 | -1.77 (0.418) | -2.02 (0.584)
  FU Phase: Week 24 | -1.70 (0.507) | -1.85 (0.616)
  FU Phase: Week 32 | -1.64 (0.616) | -1.75 (0.606)
  FU Phase: Week 40 | -1.38 (0.568) | -1.69 (0.904)
  FU Phase: Week 48: number analyzed (Participants) | 17 | 16
  FU Phase: Week 48 | -1.23 (0.527) | -1.54 (0.929)
  FU Phase: EOS | -1.26 (0.530) | -1.54 (0.929)

12. Secondary Outcome: Percentage of Participants With Change in HBsAg Levels Below/Above Different Cut-offs Over Time
Description: Percentage of participants with change in HBsAg levels below/above different cut-offs (<0.05 IU/mL, <1 U/mL, <10 IU/mL, <100 IU/mL , <1000 IU/mL) over time were reported. EOSI was the last post-baseline visit in study intervention period. EOS was the last visit in the study.
Time Frame: IP: Baseline, Weeks 1, 2, 3, 4, 8, 12, 16, 20, and EOSI (Week 24); FU Phase: FU Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, and EOS (last visit at FU Week 48)
Population: as for outcome 11
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP: Baseline: HBsAg < 0.05 IU/mL | 0 | 0
  IP: Baseline: HBsAg <1 IU/mL | 0 | 0
  IP: Baseline: HBsAg <10 IU/mL | 0 | 0
  IP: Baseline: HBsAg <100 IU/mL | 0 | 0
  IP: Baseline: HBsAg <1000 IU/mL | 38.9 | 42.1
  IP: Week 1: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 1: HBsAg <1 IU/mL | 0 | 0
  IP: Week 1: HBsAg <10 IU/mL | 0 | 0
  IP: Week 1: HBsAg <100 IU/mL | 0 | 10.5
  IP: Week 1: HBsAg <1000 IU/mL | 44.4 | 57.9
  IP: Week 2: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 2: HBsAg <1 IU/mL | 0 | 0
  IP: Week 2: HBsAg <10 IU/mL | 0 | 0
  IP: Week 2: HBsAg <100 IU/mL | 5.6 | 15.8
  IP: Week 2: HBsAg <1000 IU/mL | 38.9 | 63.2
  IP: Week 3: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 3: HBsAg <1 IU/mL | 0 | 0
  IP: Week 3: HBsAg <10 IU/mL | 0 | 0
  IP: Week 3: HBsAg <100 IU/mL | 11.1 | 15.8
  IP: Week 3: HBsAg <1000 IU/mL | 50.0 | 63.2
  IP: Week 4: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 4: HBsAg <1 IU/mL | 0 | 0
  IP: Week 4: HBsAg <10 IU/mL | 0 | 0
  IP: Week 4: HBsAg <100 IU/mL | 11.1 | 15.8
  IP: Week 4: HBsAg <1000 IU/mL | 61.1 | 73.7
  IP: Week 8: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 8: HBsAg <1 IU/mL | 0 | 0
  IP: Week 8: HBsAg <10 IU/mL | 0 | 10.5
  IP: Week 8: HBsAg <100 IU/mL | 27.8 | 42.1
  IP: Week 8: HBsAg <1000 IU/mL | 66.7 | 78.9
  IP: Week 12: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 12: HBsAg <1 IU/mL | 0 | 5.3
  IP: Week 12: HBsAg <10 IU/mL | 11.1 | 15.8
  IP: Week 12: HBsAg <100 IU/mL | 55.6 | 68.4
  IP: Week 12: HBsAg <1000 IU/mL | 100.0 | 94.7
  IP: Week 16: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 16: HBsAg <1 IU/mL | 0 | 5.3
  IP: Week 16: HBsAg <10 IU/mL | 16.7 | 21.1
  IP: Week 16: HBsAg <100 IU/mL | 83.3 | 89.5
  IP: Week 16: HBsAg <1000 IU/mL | 100.0 | 100.0
  IP: Week 20: HBsAg <0.05 IU/mL | 0 | 0
  IP: Week 20: HBsAg <1 IU/mL | 0 | 5.3
  IP: Week 20: HBsAg <10 IU/mL | 22.2 | 42.1
  IP: Week 20: HBsAg <100 IU/mL | 83.3 | 94.7
  IP: Week 20: HBsAg <1000 IU/mL | 100.0 | 100.0
  IP: EOSI (Week 24): HBsAg <0.05 IU/mL | 0 | 0
  IP: EOSI (Week 24): HBsAg <1 IU/mL | 0 | 5.3
  IP: EOSI (Week 24): HBsAg <10 IU/mL | 33.3 | 52.6
  IP: EOSI (Week 24): HBsAg <100 IU/mL | 88.9 | 94.7
  IP: EOSI (Week 24): HBsAg <1000 IU/mL | 100.0 | 100.0
  FU Phase: Week 4: HBsAg <0.05 IU/mL: number analyzed (Participants) | 6 | 7
  FU Phase: Week 4: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 4: HBsAg <1 IU/mL: number analyzed (Participants) | 6 | 7
  FU Phase: Week 4: HBsAg <1 IU/mL | 0 | 0
  FU Phase: Week 4: HBsAg <10 IU/mL: number analyzed (Participants) | 6 | 7
  FU Phase: Week 4: HBsAg <10 IU/mL | 16.7 | 57.1
  FU Phase: Week 4: HBsAg <100 IU/mL: number analyzed (Participants) | 6 | 7
  FU Phase: Week 4: HBsAg <100 IU/mL | 83.3 | 85.7
  FU Phase: Week 4: HBsAg <1000 IU/mL: number analyzed (Participants) | 6 | 7
  FU Phase: Week 4: HBsAg <1000 IU/mL | 100.0 | 100.0
  FU Phase: Week 8: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 8: HBsAg <1 IU/mL | 0 | 10.5
  FU Phase: Week 8: HBsAg <10 IU/mL | 33.3 | 52.6
  FU Phase: Week 8: HBsAg <100 IU/mL | 88.9 | 94.7
  FU Phase: Week 8: HBsAg <1000 IU/mL | 100.0 | 100.0
  FU Phase: Week 12: HBsAg <0.05 IU/mL: number analyzed (Participants) | 17 | 16
  FU Phase: Week 12: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 12: HBsAg <1 IU/mL: number analyzed (Participants) | 17 | 16
  FU Phase: Week 12: HBsAg <1 IU/mL | 0 | 0
  FU Phase: Week 12: HBsAg <10 IU/mL: number analyzed (Participants) | 17 | 16
  FU Phase: Week 12: HBsAg <10 IU/mL | 29.4 | 50.0
  FU Phase: Week 12: HBsAg <100 IU/mL: number analyzed (Participants) | 17 | 16
  FU Phase: Week 12: HBsAg <100 IU/mL | 88.2 | 93.8
  FU Phase: Week 12: HBsAg <1000 IU/mL: number analyzed (Participants) | 17 | 16
  FU Phase: Week 12: HBsAg <1000 IU/mL | 100.0 | 100.0
  FU Phase: Week 16: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 16: HBsAg <1 IU/mL | 0 | 5.3
  FU Phase: Week 16: HBsAg <10 IU/mL | 22.2 | 47.4
  FU Phase: Week 16: HBsAg <100 IU/mL | 83.3 | 94.7
  FU Phase: Week 16: HBsAg <1000 IU/mL | 100.0 | 100.0
  FU Phase: Week 20: HBsAg <0.05 IU/mL: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 20: HBsAg <1 IU/mL: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBsAg <1 IU/mL | 0 | 0
  FU Phase: Week 20: HBsAg <10 IU/mL: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBsAg <10 IU/mL | 22.2 | 52.9
  FU Phase: Week 20: HBsAg <100 IU/mL: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBsAg <100 IU/mL | 83.3 | 100.0
  FU Phase: Week 20: HBsAg <1000 IU/mL: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBsAg <1000 IU/mL | 94.4 | 100.0
  FU Phase: Week 24: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 24: HBsAg <1 IU/mL | 0 | 0
  FU Phase: Week 24: HBsAg <10 IU/mL | 16.7 | 42.1
  FU Phase: Week 24: HBsAg <100 IU/mL | 72.2 | 84.2
  FU Phase: Week 24: HBsAg <1000 IU/mL | 88.9 | 94.7
  FU Phase: Week 32: HBsAg <0.05 IU/mL | 0 | 0
  FU Phase: Week 32: HBsAg <1 IU/mL | 5.6 | 0
  FU Phase: Week 32: HBsAg <10 IU/mL | 16.7 | 26.3
  FU Phase: Week 32: HBsAg <100 IU/mL | 72.2 | 78.9
  FU Phase: Week 32: HBsAg <1000 IU/mL | 88.9 | 94.7
  FU Phase: Week 40: HBsAg <0.05 IU/mL | 0 | 5.3
  FU Phase: Week 40: HBsAg <1 IU/mL | 0 | 5.3
  FU Phase: Week 40: HBsAg <10 IU/mL | 11.1 | 15.8
  FU Phase: Week 40: HBsAg <100 IU/mL | 66.7 | 78.9
  FU Phase: Week 40: HBsAg <1000 IU/mL | 88.9 | 89.5
  FU Phase: Week 48: HBsAg <0.05 IU/mL: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBsAg <0.05 IU/mL | 0 | 5.3
  FU Phase: Week 48: HBsAg <1 IU/mL: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBsAg <1 IU/mL | 0 | 5.3
  FU Phase: Week 48: HBsAg <10 IU/mL: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBsAg <10 IU/mL | 11.8 | 15.8
  FU Phase: Week 48: HBsAg <100 IU/mL: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBsAg <100 IU/mL | 64.7 | 78.9
  FU Phase: Week 48: HBsAg <1000 IU/mL: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBsAg <1000 IU/mL | 82.4 | 89.5
  FU Phase: EOS: HBsAg <0.05 IU/mL | 0 | 5.3
  FU Phase: EOS: HBsAg <1 IU/mL | 0 | 5.3
  FU Phase: EOS: HBsAg <10 IU/mL | 11.1 | 15.8
  FU Phase: EOS: HBsAg <100 IU/mL | 66.7 | 78.9
  FU Phase: EOS: HBsAg <1000 IU/mL | 83.3 | 89.5

13. Secondary Outcome: Percentage of Participants With HBsAg Seroclearance
Description: Percentage of participants with HBsAg seroclearance were reported. Seroclearance of HBsAg was defined as a HBsAg level <lower limit of quantification (LLOQ) (0.05 IU/mL).
Time Frame: IP: Week 0 to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP | 0 | 0
  FU Phase | 0 | 5.3

14. Secondary Outcome: Percentage of Participants With HBsAg Seroconversion
Description: Percentage of participants with HBsAg seroconversion were reported. Seroconversion of HBsAg was defined as having achieved HBsAg seroclearance and appearance of anti-HBs antibodies (baseline anti-HBs antibodies <LLOQ and a post-baseline assessment >=LLOQ).
Time Frame: IP: Week 0 to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA. Here, 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure and 'n' (number analyzed) signifies number of participants analyzed for specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 17 | 19
Percentage of participants
  IP Phase | 0 | 0
  FU Phase: number analyzed (Participants) | 17 | 18
  FU Phase | 0 | 5.6

15. Secondary Outcome: Time to Achieve HBsAg Seroclearance
Description: Time to achieve HBsAg seroclearance was reported. Seroclearance of HBsAg was defined as a (quantitative) HBsAg level <LLOQ (0.05 IU/mL).
Time Frame: Week 0 up to FU Week 48 (up to Week 72)
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA. N=0 signifies that data could not be collected and analyzed as no participant had event.
Measure: Median (Full Range); unit: Days
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 0 | 1
Days |  | NA [450 to NA] — Here, 'NA' signifies that median and upper limit could not be estimated due to insufficient number of participants with events.

16. Secondary Outcome: Time to Achieve HBsAg Seroconversion
Description: Time to achieve HBsAg seroconversion were reported. Seroconversion of HBsAg was defined as having achieved HBsAg seroclearance and appearance of anti-HBs antibodies (baseline anti-HBs antibodies <LLOQ and a post-baseline assessment >=LLOQ).
Time Frame: Week 0 up to FU Week 48 (up to Week 72)
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA. Here, N=0 signifies that data could not be collected and analyzed as no participant had event.
Measure: Median (Full Range); unit: Days
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 0 | 1
Days |  | NA [505 to NA] — Here, 'NA' signifies that median and upper limit could not be estimated due to insufficient number of participants with events.

17. Secondary Outcome: Hepatitis B Virus (HBV) Deoxyribonucleic Acid (DNA) Levels Over Time
Description: HBV DNA levels over time were reported. EOSI was the last post-baseline visit in study intervention period. EOS was the last visit in the study.
Time Frame: IP: Baseline, Weeks 2, 4, 8, 12, 16, 20 and EOSI (Week 24); FU Phase: FU Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, and EOS (last visit at FU Week 48)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
log10 IU/mL
  IP: Baseline | 0.83 (0.220) | 0.80 (0.200)
  IP: Week 2 | 0.87 (0.260) | 0.72 (0.109)
  IP: Week 4 | 0.83 (0.220) | 0.85 (0.228)
  IP: Week 8 | 0.88 (0.239) | 0.82 (0.216)
  IP: Week 12 | 0.88 (0.239) | 0.82 (0.216)
  IP: Week 16 | 0.91 (0.244) | 0.82 (0.216)
  IP: Week 20 | 0.86 (0.231) | 0.80 (0.200)
  IP: EOSI (Week 24) | 0.96 (0.281) | 0.77 (0.179)
  FU Phase: Week 4 | 0.83 (0.220) | 0.90 (0.288)
  FU Phase: Week 8 | 0.83 (0.220) | 0.80 (0.200)
  FU Phase: Week 12: number analyzed (Participants) | 17 | 18
  FU Phase: Week 12 | 0.93 (0.257) | 0.91 (0.244)
  FU Phase: Week 16 | 0.78 (0.183) | 0.85 (0.228)
  FU Phase: Week 20: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20 | 0.86 (0.231) | 0.90 (0.242)
  FU Phase: Week 24 | 0.86 (0.231) | 0.87 (0.236)
  FU Phase: Week 32 | 0.88 (0.239) | 0.75 (0.150)
  FU Phase: Week 40 | 0.91 (0.244) | 0.85 (0.228)
  FU Phase: Week 48: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48 | 0.84 (0.224) | 0.82 (0.216)
  FU Phase: EOS | 0.83 (0.220) | 0.82 (0.216)

18. Secondary Outcome: Percentage of Participants With Hepatitis B Virus Deoxyribonucleic Acid (HBV DNA) Level Below/Above Different Cut-offs Over Time
Description: Percentage of participants with HBV DNA level below/above different cut-offs over time were reported. HBV DNA cut offs: <LLOQ target detected (TD): that is, traces of HBV DNA were detected/found but were too low to be quantified; <LLOQ target not detected (TND): that is, no traces of HBV DNA were detected/found. EOSI was the last post-baseline visit in study intervention period. EOS was the last visit in the study. The LLOQ for HBV DNA was 20 IU/mL. As indicated in the data table, the sum of percentage values of each sub-categories within the specific timepoints "IP: Week 2" and "FU Phase: Week 4", shows a slight deviation from 100% due to rounding.
Time Frame: IP: Baseline, Weeks 2, 4, 8, 12, 16, 20, and EOSI (Week 24); FU Phase: FU Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, and EOS (last visit at FU Week 48)
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP: Baseline: HBV DNA < LLOQ TND | 72.2 | 78.9
  IP: Baseline: HBV DNA < LLOQ TD | 27.8 | 21.1
  IP: Week 2: HBV DNA < LLOQ TND | 66.7 | 94.7
  IP: Week 2: HBV DNA < LLOQ TD | 27.8 | 5.3
  IP: Week 2: HBV DNA > LLOQ | 5.6 | 0
  IP: Week 4: HBV DNA < LLOQ TND | 72.2 | 68.4
  IP: Week 4: HBV DNA < LLOQ TD | 27.8 | 31.6
  IP: Week 8: HBV DNA < LLOQ TND | 61.1 | 73.7
  IP: Week 8: HBV DNA < LLOQ TD | 38.9 | 26.3
  IP: Week 12: HBV DNA < LLOQ TND | 61.1 | 73.7
  IP: Week 12: HBV DNA < LLOQ TD | 38.9 | 26.3
  IP: Week 16: HBV DNA <LLOQ TND | 55.6 | 73.7
  IP: Week 16: HBV DNA <LLOQ TD | 44.4 | 26.3
  IP: Week 20: HBV DNA <LLOQ TND | 66.7 | 78.9
  IP: Week 20: HBV DNA <LLOQ TD | 33.3 | 21.1
  IP: EOSI(Week 24): HBV DNA <LLOQ TND | 50.0 | 84.2
  IP: EOSI(Week 24): HBV DNA <LLOQ TD | 38.9 | 15.8
  IP: EOSI(Week 24): HBV DNA > LLOQ | 11.1 | 0
  FU Phase: Week 4: HBV DNA <LLOQ TND | 72.2 | 63.2
  FU Phase: Week 4: HBV DNA <LLOQ TD | 27.8 | 31.6
  FU Phase: Week 4: HBV DNA > LLOQ | 0 | 5.3
  FU Phase: Week 8: HBV DNA <LLOQ TND | 72.2 | 78.9
  FU Phase: Week 8: HBV DNA <LLOQ TD | 27.8 | 21.1
  FU Phase: Week 12: HBV DNA <LLOQ TND: number analyzed (Participants) | 17 | 18
  FU Phase: Week 12: HBV DNA <LLOQ TND | 52.9 | 55.6
  FU Phase: Week 12: HBV DNA <LLOQ TD: number analyzed (Participants) | 17 | 18
  FU Phase: Week 12: HBV DNA <LLOQ TD | 41.2 | 44.4
  FU Phase: Week 12: HBV DNA > LLOQ | 5.9 | 0
  FU Phase: Week 16: HBV DNA <LLOQ TND | 83.3 | 68.4
  FU Phase: Week 16: HBV DNA <LLOQ TD | 16.7 | 31.6
  FU Phase: Week 20: HBV DNA <LLOQ TND: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBV DNA <LLOQ TND | 66.7 | 58.8
  FU Phase: Week 20: HBV DNA <LLOQ TD: number analyzed (Participants) | 18 | 17
  FU Phase: Week 20: HBV DNA <LLOQ TD | 33.3 | 41.2
  FU Phase: Week 24: HBV DNA <LLOQ TND | 66.7 | 63.2
  FU Phase: Week 24: HBV DNA <LLOQ TD | 33.3 | 36.8
  FU Phase: Week 32: HBV DNA <LLOQ TND | 61.1 | 89.5
  FU Phase: Week 32: HBV DNA <LLOQ TD | 38.9 | 10.5
  FU Phase: Week 40: HBV DNA <LLOQ TND | 55.6 | 68.4
  FU Phase: Week 40: HBV DNA <LLOQ TD | 44.4 | 31.6
  FU Phase: Week 48: HBV DNA <LLOQ TND: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBV DNA <LLOQ TND | 70.6 | 73.7
  FU Phase: Week 48: HBV DNA <LLOQ TD: number analyzed (Participants) | 17 | 19
  FU Phase: Week 48: HBV DNA <LLOQ TD | 29.4 | 26.3
  FU Phase: EOS: HBV DNA <LLOQ TND | 72.2 | 73.7
  FU Phase: EOS: HBV DNA <LLOQ TD | 27.8 | 26.3

19. Secondary Outcome: Percentage of Participants With Hepatitis B e Antigen (HBeAg) Level Below/Above Different Cut-offs Over Time
Description: Percentage of participants with HBeAg level below/above different cut-offs over time were reported. HBeAg cut-offs: <LLOQ (0.11 IU/mL). EOSI was the last post-baseline visit in study intervention period. EOS was the last visit in the study.
Time Frame: IP: Baseline, Weeks 2, 4, 8, 12, 20, and EOSI (Week 24); FU Phase: FU Weeks 12, 16, 20, 24, 32, 40, 48, and EOS (last visit at FU Week 48)
Population: FAS included all participants who were randomly assigned to an intervention arm in this ISA and received at least 1 dose of study intervention within this ISA. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified timepoint. Here, n=0 signifies no participant was analyzed at specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP: Baseline | 100.0 | 94.7
  IP: Week 2: number analyzed (Participants) | 0 | 1
  IP: Week 2 |  | 100
  IP: Week 4: number analyzed (Participants) | 0 | 1
  IP: Week 4 |  | 100.0
  IP: Week 8: number analyzed (Participants) | 0 | 1
  IP: Week 8 |  | 100.0
  IP: Week 12 | 100.0 | 100.0
  IP: Week 20: number analyzed (Participants) | 0 | 1
  IP: Week 20 |  | 100.0
  IP: EOSI (Week 24) | 100.0 | 100.0
  FU Phase: Week 12: number analyzed (Participants) | 16 | 16
  FU Phase: Week 12 | 100.0 | 100.0
  FU Phase: Week 16: number analyzed (Participants) | 0 | 1
  FU Phase: Week 16 |  | 100.0
  FU Phase: Week 24: number analyzed (Participants) | 18 | 18
  FU Phase: Week 24 | 100.0 | 100.0
  FU Phase: Week 32: number analyzed (Participants) | 0 | 1
  FU Phase: Week 32 |  | 100.0
  FU Phase: Week 40: number analyzed (Participants) | 1 | 0
  FU Phase: Week 40 | 100.0 |
  FU Phase: Week 48: number analyzed (Participants) | 17 | 17
  FU Phase: Week 48 | 94.1 | 100.0
  FU Phase: EOS | 94.4 | 100.0

20. Secondary Outcome: Percentage of Participants With Virologic Breakthrough
Description: Percentage of participants with virologic breakthrough (confirmed on-treatment HBV DNA increase by >1 log10 IU/mL from nadir in participants who did not have on-treatment HBV DNA level below LLOQ or a confirmed on-treatment HBV DNA level >200 IU/mL in participants who had on-treatment HBV DNA level below LLOQ) were reported.
Time Frame: IP: Week 0 to Week 24; FU Phase: FU Week 1 up to FU Week 48
Population: FAS included all participants who were randomly assigned to an intervention arm in this intervention-specific appendix (ISA) and received at least 1 dose of study intervention within this ISA.
Measure: Number; unit: Percentage of participants
Arm/Group | JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | JNJ-3989 + Nivolumab (3 Infusions) + NA
Number analyzed (Participants) | 18 | 19
Percentage of participants
  IP | 0 | 0
  FU Phase | 0 | 0

ADVERSE EVENTS:
Time Frame: IP: Week 0 up to Week 24; FU Phase: FU Week 1 up to FU Week 48
Description: Safety analysis set included all subjects who received at least 1 dose of study intervention within this ISA.
Groups:
- IP: JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA: In intervention phase (IP), participants received a loading dose of JNJ-3989 200 milligrams (mg) as subcutaneous (SC) injection once weekly (QW) for first 4 weeks starting from Week 0 up to Week 3 followed by single dose once every 4 weeks (Q4W) from Week 4 up to Week 24. At Week 16, participants received a single dose of nivolumab 0.3 mg/kg as intravenous (IV) infusion. Participants also received NA (either tenofovir disoproxil 245 mg or tenofovir alafenamide [TAF] 25 mg or entecavir [ETV] 0.5 mg) tablet orally once daily (QD) from Week 0 up to Week 24.
- IP: JNJ-3989 + Nivolumab (3 Infusions) + NA: In IP, participants received a loading dose of JNJ-3989 200 mg as SC injection QW for first 4 weeks starting from Week 0 up to Week 3 followed by single dose Q4W from Week 4 up to Week 24. At Weeks 16, 20 and 24, participants received of nivolumab 0.3 mg/kg as IV infusion. Participants also received NA (either tenofovir disoproxil 245 mg or TAF 25 mg or ETV 0.5 mg) tablet orally QD from Week 0 up to Week 24.
- FU: JNJ-3989 + Nivolumab (1 Infusion) + NA; FU: JNJ-3989 + Nivolumab (3 Infusions) + NA: After Week 24, participants were followed up for safety for 48 weeks during which they continued to receive NA (tenofovir disoproxil 245 mg or TAF 25 mg or ETV 0.5 mg) tablet orally QD up to FU Week 48 (up to Week 72).
Arm/Group | IP: JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA | IP: JNJ-3989 + Nivolumab (3 Infusions) + NA | FU: JNJ-3989 + Nivolumab (1 Infusion) + NA | FU: JNJ-3989 + Nivolumab (3 Infusions) + NA
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 6/18 | 12/19 | 8/18 | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IP: JNJ-73763989 (JNJ-3989) + Nivolumab (1 Infusion) + NA (N=18) | IP: JNJ-3989 + Nivolumab (3 Infusions) + NA (N=19) | FU: JNJ-3989 + Nivolumab (1 Infusion) + NA (N=18) | FU: JNJ-3989 + Nivolumab (3 Infusions) + NA (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Conjunctival Haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0
Injection Site Erythema (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0
Candida Infection (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 3 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 1 | 0
Laryngopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1
Amylase Increased (Investigations) | 0 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervical Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Cyst (Renal and urinary disorders) | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Intermenstrual Bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Per protocol amendment 2 (28 Mar 2023), due to difficulties in recruitment, further participants enrollment was stopped. Hence, pharmacokinetic assessments were not performed due to change in planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT05275023/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT05275023/SAP_001.pdf